CLINICAL TRIAL: NCT07153744
Title: Efficacy and Safety of Shexiang Baoxin Pill(MUSKARDIA) in the Treatment of Acute Myocardial Infarction: A Prospective, Multicenter, Pragmatic Randomized Controlled Real-World Study
Brief Title: Efficacy and Safety of Shexiang Baoxin Pill(MUSKARDIA) in the Treatment of Acute Myocardial Infarction
Acronym: MUST Ⅱ
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Hutchison Pharmaceuticals Limited (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other); Huashan Hospital (Other); Shanghai 10th People's Hospital (Other); Shanghai 6th People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai East Hospital (Other); Longhua Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Affiliated Hospital of Jiangsu University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First People's Hospital of Lianyungang (Other); Huai'an First People's Hospital (Other); Sir Run Run Shaw Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital of Ningbo University (Network); Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Weihai Municipal Hospital (Other); Weifang People's Hospital (Other); Rizhao People's Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Jining First People's Hospital (Other); Linyi People's Hospital (Other); Xiangya Hospital of Central South University (Other); Second Xiangya Hospital of Central South University (Other); Yueyang Central Hospital (Other); The First Affiliated Hospital of University of South China (Other); The Central Hospital of Shaoyang (Unknown); The First People's Hospital of Changde City (Other); Wuxi People's Hospital (Other); Jinhua Central Hospital (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other); Shuguang Hospital of Shanghai University of Traditional Chinese Medicine (Unknown); Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other); ZhuZhou Central Hospital (Other); First People's Hospital of Chenzhou (Other); People's Hospital of Quzhou (Other); Xuzhou New Health Hospital (Unknown); Taizhou Enze Medical Center Group (Other); Beijing Chao Yang Hospital (Other); Civil Aviation General Hospital (Other); Xuanwu Hospital, Beijing (Other); Beijing Friendship Hospital (Other); Peking University People's Hospital (Other); Beijing Electric Power Hospital (Other); Renmin Hospital of Wuhan University (Other); Wuhan No.1 Hospital (Other); Jingzhou Central Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Ansteel Group General Hospital (Unknown); General Hospital of Fuxin Mining Industry Group of Liaoning Health Industry Group (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Huaihe Hospital of Henan University (Other); Zhoukou Central Hospital (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other); First Affiliated Hospital of Nanyang Medical College (Other); Jiaozuo Second People's Hospital (Unknown); Anyang Area Hospital of Puyang City (Unknown); Shijiazhuang People's Hospital (Other); Cangzhou Central Hospital (Other); The First Hospital of Hebei Medical University (Other); Handan Central Hospital (Other); The People's Hospital of Langfang City (Unknown); Xingtai Central Hospital (Unknown); North China University of Science and Technology (Other); The First Affiliated Hospital of Anhui Medical University (Other); the First Hospital of Anhui University of Science and Technology (Unknown); Chaohu Hospital of Anhui Medical University (Other); Tongling People's Hospital (Other Government); Huang Shan People's Hospital (Other); Huaibei Miners General Hospital (Unknown); The Second Affiliated Hospital of Fujian Medical University (Other); Changzhi Medical College (Other); LinFen People's Hospital (Unknown); Shanxi Cardiovascular Hospital (Other); Dazhou First People's Hospital (Unknown); The Affiliated Hospital Of Southwest Medical University (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); Yangchun People's Hospital (Unknown); Shaoguan People's Hospital (Unknown); Guilin People's Hospital (Unknown); The First Affiliated Hospital of Nanchang University (Other); Ji'an Central People's Hospital (Unknown); Jiangxi Provincial People's Hopital (Other); People's Hospital of Chongqing (Other); Ankang Central Hospital (Other); Xiangyang Central Hospital (Other); Tianjin Third Central Hospital (Other); General Hospital of Ningxia Medical University (Other); The Second Affiliated Hospital of Hainan Medical University (Other); Lanzhou University Second Hospital (Other); Jilin Province People's Hospital (Unknown); Inner Mongolia Autonomous Region People's Hospital (Unknown); Yan'an Hospital of Kunming City (Unknown); The People's Hospital of Jizhou District, Tianjin (Unknown); The Southwest Hospital of Army Medical University (Unknown); The First People's Hospital of Nanning (Unknown); The People' s Hospital of Jiangmen (Unknown); The second People's Hospital of Guiyang (Unknown); The Third People's Hospital of Chengdu (Other); The Tirst People's Hospital of Mianyang (Unknown); First Affiliated Hospital of Fujian Medical University (Other); The First People's Hospital of Chu Zhou (Unknown); Xuancheng people's hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPE202501
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Acute Myocardial Infarction (AMI); Percutaneous Coronary Intervention (PCI)
Keywords: Acute Myocardial Infarction; AMI; Percutaneous Coronary Intervention; PCI; Shexiang Baoxin Pill; MUSKARDIA; Shexiang Baoxin Pill(MUSKARDIA); SBP
MeSH Terms: interventions — Aspirin; Adrenergic beta-Antagonists; Cholesterol; Diet; Educational Status; Exercise; shexiang baoxin

STUDY DESIGN:
Intervention Model Description: Stratified block randomization by center was performed using a computer-generated random sequence to allocate patients to the Shexiang Baoxin Pill group and the conventional treatment group at a ratio of 2:1.
  Patients in the Shexiang Baoxin Pill group initiated treatment immediately after randomization. They received 2-4 pills of Shexiang Baoxin Pill preoperatively before PCI, followed by a maintenance dose of 2-4 pills orally three times daily (TID) with warm water for 12 months postoperatively, concurrently with standard guideline-directed therapy.
  Patients in the conventional treatment group will receive standard treatment in accordance with guidelines and consensuses after surgery, and this will last for 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Shexiang Baoxin Pill Group (Experimental): Patients in the Shexiang Baoxin Pill group initiated treatment immediately after randomization. They received 2-4 pills of Shexiang Baoxin Pill preoperatively before PCI, followed by a maintenance dose of 2-4 pills orally three times daily (TID) with warm water for 12 months postoperatively, concurrently with standard guideline-directed therapy.
  Interventions: Drug: Shexiang Baoxin Pill
- the Conventional Treatment Group (Active Comparator): Patients in the conventional treatment group will receive standard treatment in accordance with guidelines and consensuses after surgery, and this will last for 12 months.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Patients in the Shexiang Baoxin Pill(MUSKARDI) group initiated treatment immediately after randomization. They received 2-4 pills of Shexiang Baoxin Pill preoperatively before PCI, followed by a maintenance dose of 2-4 pills orally three times daily (TID) with warm water for 12 months postoperatively, concurrently with standard guideline-directed therapy.
  Other Names: standard guideline-directed therapy; ABCDE; Antiplatelet; Beta-blocker; Cholesterol; Diet & Diabetes; Education & Exercise
  Arms: the Conventional Treatment Group
Drug: Shexiang Baoxin Pill — Patients in the Shexiang Baoxin Pill group initiated treatment immediately after randomization. They received 2-4 pills of Shexiang Baoxin Pill preoperatively before PCI, followed by a maintenance dose of 2-4 pills orally three times daily (TID) with warm water for 12 months postoperatively, concurrently with standard guideline-directed therapy.
  Arms: the Shexiang Baoxin Pill Group

SUMMARY:
This study aims to evaluate the value of Shexiang Baoxin Pill (MUSKARDIA) in patients with acute myocardial infarction (AMI) through a prospective, multicenter, pragmatic randomized controlled real-world study. It seeks to validate its efficacy in reducing cardiovascular event risk during the peri-PCI period, as well as its effects on cardiac function, quality of life , and relevant biomarkers. Through this research, we expect to provide higher-quality evidence for the application of SBP in AMI patients undergoing PCI, thereby further optimizing comprehensive treatment strategies for AMI.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, regardless of gender
* In accordance with the 2023 ESC Guidelines for the Management of Acute Coronary Syndromes , meeting the diagnostic criteria for acute myocardial infarction, including typical chest pain lasting for ≥20 minutes, electrocardiographic manifestations of ST-segment elevation (STEMI) or non-ST-segment elevation myocardial infarction (NSTEMI), and serum high-sensitivity troponin (hs-cTn) levels exceeding the 99th percentile of the upper reference limit at least once with dynamic changes
* Presenting for treatment within <24 hours of symptom onset and scheduled to undergo PCI
* The patient or their guardian has signed the informed consent form

Exclusion Criteria:

* Having contraindications to PCI treatment
* Being allergic to Shexiang Baoxin Pills, unable to tolerate them, or having other conditions that prevent completion of the trial drug administration
* Being pregnant, planning to become pregnant, or breastfeeding women
* Having participated in other clinical studies within 3 months
* Being deemed unsuitable for inclusion in this study by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9588 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular and cerebrovascular events (MACE) | 1 year after PCI
  Cumulative incidence of MACE events at 1 year from the start of randomization. MACE events include cardiac death, non-fatal myocardial infarction, non-fatal stroke, re-hospitalization for angina pectoris, and unplanned revascularization.

SECONDARY OUTCOMES:
Incidence of non-fatal myocardial infarction | 1 year after PCI
Incidence of non-fatal stroke | 1 year after PCI
Rehospitalization rate due to angina pectoris | 1 year after PCI
Rate of unplanned revascularization | 1 year after PCI
Cardiac mortality rate | 1 year after PCI
Rehospitalization rate due to heart failure | 1 year after PCI
All-cause mortality rate | 1 year after PCI
  All-cause mortality rate: including cardiac and non-cardiac deaths
Seattle Angina Questionnaire score | 1 year after PCI
EQ-5D-5L scale | 1 year after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: National Universal Health Security Information Platform - Medical Research Registration and Filing Information System — https://www.medicalresearch.org.cn/clinicalResearch/researchInfo?id=7e01c957-3c11-4313-95f7-2b9468af2913